CLINICAL TRIAL: NCT05706675
Title: Specialized Pro-resolving Mediators (SPM) as Biomarkers of Periodontal Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Zahi BADRAN, Professor, University of Sharjah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: REC-22-02-28-02-S
Record Dates: First submitted 2023-01-21; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Inflammation; Periodontitis
MeSH Terms: conditions — Inflammation; Periodontitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Periodontitis patients that will be treatyed with Non surgical Periodontal Therapy
  Interventions: Procedure: Non surgical periodontal therapy
- Control (No Intervention): Periodontally healthy patients

INTERVENTIONS:
Procedure: Non surgical periodontal therapy — Manual root planning+Ultrasonic subgingival debridement
  Arms: Experimental

SUMMARY:
Periodontal diseases are a public health burden in all countries. Hence, Periodontitis is the sixth-most prevalent disease in the world, the most common bone diseases in human and the primary cause for tooth loss in adults leading to significant economic and medical consequences. All disease biomarkers could help to stratify the general population with those at high risk of periodontitis and to enroll them in a rigorous prevention program. Advanced periodontitis has been shown to reduce the quality of life of patients and developing novel biological monitoring protocols will reduce the prevalence of advanced forms of the disease.

There are alot of research explaining the different types of inflammatory mediators that could be found in periodontitis patients. But there are a few research have been talking about lipoxin A4 as an inflammatory biomarker that could detect the effect of non surgical periodontal therapy effect on the periodontal health.

And the aim of the study is to assess the effect of this non surgical periodontal therapy on the periodontal health by assessing the concentration of this biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Control group : Patients diagnosed as periodontally healthy
* Test group:

  * Patients diagnosed with generalized periodontitis (Stage 3/4, Grade a,b or c).
  * Having at least 15 remaining teeth.
  * Mentally able to understand the communication and to express an informed consent

Exclusion Criteria:

* Systemic diseases with known effect on periodontal health
* Antibiotics/Anti-inflammatory drugs taken in the last month
* Women with suspected/known pregnancy, or taking any hormone-based treatment
* Patients suffering from Xerostomia.
* Patients smoking more than 20 cig/day.
* Previous periodontal therapy in the last 3-6 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Lipoxin A4 | 2 months
  Gingival crevicular fluid concentration

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Zahi Badran, Phd, Study Director — University of Sharjah
Locations (1):
- University Dental Hospital Sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No